CLINICAL TRIAL: NCT00761761
Title: Sensoril® (Ashwagandha) - A Standardized Extract From a Medicinal Plant - (Withania Somnifera) for Cognitive Enhancement in Persons With Bipolar Disorder: A Parallel Group, Randomized Double Blind, and Placebo Controlled Study
Brief Title: Sensoril(Ashwaganhda)for Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, K.N. Roy Chengappa, Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Chengappa Sensoril; Univ.Pitts IRB# PRO08060267
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Results first posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Bipolar I Disorder; Bipolar II Disorder; Bipolar Disorder NOS
Keywords: Sensoril; Bipolar Illness; Cognitive enhancement
MeSH Terms: conditions — Bipolar Disorder | interventions — Ashwagandha; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1- Sensoril (Ashwagandha) (Experimental): Sensoril (Ashwagandha) will be administered using random assignment at a dose of 250 mg/day, increasing to a dose of 500 mg/day by the second week.
  Interventions: Drug: Sensoril
- 2 - Placebo (Placebo Comparator): Placebo will be administered using random assignment at a dose of 250 mg/day, increasing to a dose of 500 mg/day by the second week.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sensoril
  Other Names: Ashwagandha
  Arms: 1- Sensoril (Ashwagandha)
Other: Placebo
  Other Names: Sugar Pill
  Arms: 2 - Placebo

SUMMARY:
The investigators hypothesis is that oral Sensoril® (as compared to placebo) will enhance cognitive abilities (specifically measures of attention, executive function, working memory, and visuospatial ability) in persons with bipolar disorder. Secondarily, the investigators hypothesize there will be secondary improvements in residual mood/anxiety symptoms, and metabolic indices, if impaired (fasting blood glucose and lipids).

The investigators aim to test these hypotheses by conducting a randomized, placebo controlled, add on treatment trial of Sensoril® (added to existing mood stabilizer treatment) recruiting 60 subjects with DSM IV-TR bipolar disorder for a period of 8 weeks. Measures of cognition, psychopathology and laboratory indices will be utilized for evaluating primary and secondary outcomes, along with safety assessments.

DETAILED DESCRIPTION:
OBJECTIVE:

To evaluate if Sensoril® treatment of persons with bipolar illness will improve their cognitive performance and if it will improve residual mood/anxiety symptoms and impaired metabolic indices.

RESEARCH PLAN:

We will conduct a randomized, placebo controlled, add on treatment trial of Sensoril® (added to ongoing prescribed pharmacological mood stabilizer) for a period of 8 weeks. Measures of cognition, psychopathology and laboratory indices will be utilized for evaluating primary and secondary outcomes, along with safety assessments.

METHODS:

Up to Seventy-six subjects with DSM IV bipolar I disorder will be recruited from Western Psychiatric Institute and Clinic. Using a 1:1 randomization, subjects who sign an informed consent document will be randomized to receive Sensoril® or placebo.

It is expected that 16 of the 76 subjects may not meet inclusion/exclusion criteria, leaving 60 consenting adults (18 to 65 years) with DSM IV-TR Bipolar Disorder who will be assessed for euthymia (Young Mania Rating Scale Score of less than or equal to 10, Montgomery Asberg Depression Rating Scale Score of less than or equal to 10) over the period of 4 weeks while receiving stable doses of their current mood stabilizer. They will also be assessed for cognitive dysfunction (attention/executive function, immediate and declarative memory, psychomotor performance) using Cogtest - a proprietary neuropsychological battery of tests. These subjects will be characterized for normal pre-morbid IQ, no ECT treatment in past 6 months, no alcohol or substance dependence in past 6 months, mini-mental state score of 23 or more.

Sensoril® (or placebo) will be administered using random assignment at a dose of 250mg/day, increasing to a dose of 500mg/day by the second week. The dose of 500mg (or 250mg if tolerability is an issue) will be continued fora total of 8 weeks. Sensoril® is not known to have interactions with psychotropic drugs, but mood-stabilizer levels will be monitored at the beginning and end of the study. The principal investigator has worked with a New Jersey based company (Natreon, Inc.) to obtain an IND from the FDA for Sensoril® treatment of cognitive dysfunction in persons with Bipolar disorder (IND #102616).

Standard psychopathology rating scales will be administered to evaluate impact if any on residual symptoms of bipolar disorder. Laboratory indices (glucose/lipids) will be evaluated at baseline and end of study. Safety will be assessed through a comprehensive health assessment, including medical history, and evaluation of laboratory measures. Any adverse effects will be assessed by asking questions at each visit, and if necessary, follow up via telephone contact or bringing subjects in for assessments outside the scheduled visits.

SIGNIFICANCE:

Cognitive dysfunction can seriously hinder improved functional outcomes in persons with bipolar disorder. If this short term intervention with Sensoril® shows promise, more definitive studies using adequate powered sample sizes, and of longer duration can be conducted. If improvements in cognitive problems are linked to improved functional outcomes using such supplemental treatments, an important therapeutic milestone in bipolar disorder will have been achieved.

ELIGIBILITY:
Inclusion Criteria:

* DSMIV-TR diagnosis of Bipolar Disorder
* Ages 18 to 65
* Men or Women
* 8th grade education or greater
* Able to provide competent written informed consent
* Current main mood stabilizer and mood status (YMRS and MADRS scores less than or equal to 10) are stable for greater than or equal to 4 weeks by history.

Exclusion Criteria:

* Medically unstable conditions
* Known allergy to Sensoril® (or Ashwagandha)
* Current cognitive decline is attributable to a diagnosis of dementia or other neurological disorder
* Pregnant or lactating women
* Mini-mental score (MMSE) less than or equal to 23
* Currently receiving donepezil, rivastigamine, or galatamine, or memantine or any marketed agent for slowing memory loss in dementia
* Abnormal clinical thyroid status
* Currently (or within past 2 weeks) receiving St. John's Wort, Gingko or Omega-3

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K. N. Roy Chengappa, MD, Principal Investigator — Western Psychiatric Institute and Clinic
Locations (2):
- United States (2):
  - Western Psychiatric Institute and Clinic University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Chengappa KN, Bowie CR, Schlicht PJ, Fleet D, Brar JS, Jindal R. Randomized placebo-controlled adjunctive study of an extract of withania somnifera for cognitive dysfunction in bipolar disorder. J Clin Psychiatry. 2013 Nov;74(11):1076-83. doi: 10.4088/JCP.13m08413. PMID 24330893
- See also: Connect to NARSAD list of active research studies — http://www.narsad.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Sensoril Ashwagandha -1: Sensoril(Ashwagandha)
  Sensoril: Sensoril® (or placebo) will be administered using random assignment at a dose of 250mg/day, increasing to a dose of 500mg/day by the second week. The dose of 500mg (or 250mg if tolerability is an issue) will be continued for a total of 8 weeks.
- Placebo - 2: Placebo
  Sensoril: Sensoril® (or placebo) will be administered using random assignment at a dose of 250mg/day, increasing to a dose of 500mg/day by the second week. The dose of 500mg (or 250mg if tolerability is an issue) will be continued for a total of 8 weeks.
Period: Overall Study
Arm/Group | Sensoril Ashwagandha -1 | Placebo - 2
Started | 30 | 30
Completed | 24 | 29
Not Completed | 6 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sensoril: Sensoril(Ashwagandha)
  Sensoril: Sensoril® will be administered using random assignment at a dose of 250mg/day, increasing to a dose of 500mg/day by the second week. The dose of 500mg (or 250mg if tolerability is an issue) will be continued for a total of 8 weeks.
- Placebo: Placebo
  Placebo will be administered using random assignment at a dose of 250 mg/day, increasing to a dose of 500 mg/day by the second week and will be continued for a total of 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Sensoril | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (10.38) | 45.93 (10.40) | 46.42 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 17 | 20 | 37
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Digit-Span Score at 8 Weeks
Description: Cognition was assessed using tests developed by The Cognition Group-(TCG); London, UK; and Delaware, USA. Testing procedures and consistency was assured by the same staff-patient dyad, and a TCG staff person had previously trained the research staff (Chengappa et al, 2012). A comprehensive cognitive battery was assessed. Details of these cognitive tests are available at http://www.cogtest.com, and are also described in other studies (Harvey et al, 2007, Lindenmayer et al, 2011, Chengappa et al, 2012). However, the results for Digit span which assesses short term or working memory are presented.
  The raw scores for "digit span" ranges from a minimum of 2 to a maximum of 8. The Digit Span test measures working memory and the longer the span the better the cognition therefore the higher score is the better outcome.
Time Frame: 8 week treatment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Sensoril: Sensoril(Ashwagandha)
  Sensoril: Sensoril® (or placebo) will be administered using random assignment at a dose of 250mg/day, increasing to a dose of 500mg/day by the second week. The dose of 500mg (or 250mg if tolerability is an issue) will be continued for a total of 8 weeks.
- Placebo: Placebo
  Sensoril: Sensoril® (or placebo) will be administered using random assignment at a dose of 250mg/day, increasing to a dose of 500mg/day by the second week. The dose of 500mg (or 250mg if tolerability is an issue) will be continued for a total of 8 weeks.
Arm/Group | Sensoril | Placebo
Number analyzed (Participants) | 24 | 29
units on a scale | 0.73 (0.19) | 0.17 (0.18)

2. Secondary Outcome: Sensoril® Treatment Will Secondarily Improve Any Residual Depressive Symptoms
Description: Depressive symptoms were measured using the Montgomery-Asberg Depression Rating Scale (MADRS). Minimum score = 0, Maximum score = 60. Higher scores on MADRS indicate worse functioning.
Time Frame: Baseline and 8 week treatment
Population: Stable Bipolar patients
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sensoril Ashwagandha -1 | Placebo - 2
Number analyzed (Participants) | 29 | 30
units on a scale
  Baseline | 6.2 (3.6) | 4.8 (3.6)
  8 weeks | 4.8 (4.3) | 4.1 (4.7)

3. Secondary Outcome: Sensoril Treatment Will Secondarily Improve Any Residual Symptoms of Mania.
Description: Manic symptoms were measured using the Young Mania Rating Scale (YMRS). Minimum score = 0, Maximum score = 60. Higher scores on YMRS indicate worse functioning.
Time Frame: Baseline and 8 weeks treatment
Population: Stable Bipolar Patients
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sensoril Ashwagandha -1 | Placebo - 2
Number analyzed (Participants) | 29 | 30
units on a scale
  Baseline | 3.9 (2.3) | 3.7 (2.2)
  8 Weeks | 2.8 (2.4) | 3.2 (2.7)

4. Secondary Outcome: Sensoril Treatment Will Secondarily Improve Any Residual Anxiety Symptoms
Description: Symptoms of anxiety were measured using the Hamilton Anxiety Rating Scale (HARS). Minimum score = 0, Maximum score = 60. Higher scores on HARS indicate worse functioning
Time Frame: Baseline and 8 week treatment
Population: Stable Bipolar Patients
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sensoril Ashwagandha -1 | Placebo - 2
Number analyzed (Participants) | 29 | 30
units on a scale
  Baseline | 3.8 (4.5) | 5.3 (5.6)
  8 weeks | 3.2 (5.6) | 4.1 (5.8)

ADVERSE EVENTS:
Arm/Group | Sensoril | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 5/30 | 1/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensoril (N=30) | Placebo (N=30)
diarrhea (Gastrointestinal disorders) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No